CLINICAL TRIAL: NCT03702946
Title: Effect of Oxytocin Infusion on Reducing the Blood Loss During Abdominal Myomectomy: A Randomized Controlled Trial
Brief Title: Oxytocin Infusion and Abdominal Myomectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Armed Forces Hospital, Pakistan (Other)
Responsible Party: Principal Investigator, arshad khushdil, Assistant professor, Armed Forces Hospital, Pakistan
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: OXYTOCIN
Record Dates: First submitted 2018-10-06; First posted 2018-10-11 (Actual); Last update posted 2018-10-11 (Actual); Status verified 2018-10

CONDITIONS: Oxytocin and Abdominal Myomectomy
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental)
  Interventions: Other: oxytocin in abdominal myomectomy
- control group (No Intervention)

INTERVENTIONS:
Other: oxytocin in abdominal myomectomy — Women were divided into two groups randomly. In the study group 30 Units of oxytocin in 1000 ml normal saline were given during surgery, at the rate of 15units/hour. In control group, pure normal saline was given
  Arms: study group

SUMMARY:
Objective:To compare oxytocin infusion with control, in patients undergoing abdominal myomectomy in terms of mean blood loss.

Design: Single blinded randomized control trial Setting: Obstetrics and Gynecology Department, Military Hospital, Rawalpindi Population: 60 women of ASA class I-II, with intramural fibroids, candidate for elective abdominal myomectomy.

Methods: Women were divided into two groups randomly. In the study group 30 Units of oxytocin in 1000 ml normal saline were given during surgery, at the rate of 15units/hour. In control group, pure normal saline was given.

Main outcome measure: Intra-operative blood loss

ELIGIBILITY:
Inclusion Criteria:

1. women of ASA class I-II with intramural fibroids,
2. women planned to undergo elective abdominal myomectomy

Exclusion Criteria:

1. Women with hemoglobin (Hb) < 10g/dl
2. Women with any respiratory or cardiovascular disease.

Ages: 25 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2017-07-15 (Actual); Primary Completion 2018-01-15 (Actual); Study Completion 2018-01-15 (Actual)

PRIMARY OUTCOMES:
Intra-operative blood loss | during the surgical procedure
  average intra operative blood loss was measured

CONTACTS AND LOCATIONS:
Locations (2):
- Pakistan (2):
  - Department of Pediatrics, Rawalpindi, Punjab Province
  - Military Hospital, Rawalpindi, Punjab Province

IPD SHARING:
Plan to Share IPD: No